CLINICAL TRIAL: NCT00665119
Title: Effects of Remifentanil on Breathing Pattern, Respiratory Effort and Gas Exchange in Mechanically Ventilated Patients.
Brief Title: Effects of Remifentanil on Respiratory Function in Mechanically Ventilated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Natalini Giuseppe, FPoliambulanza
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FP-TIP-01
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Respiratory Insufficiency; Respiration, Artificial; Conscious Sedation
Keywords: Respiratory Insufficiency; Respiration, Artificial; Remifentanil; Respiratory Mechanics; Work of Breathing
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): Any patient alternatively receive both remifentanil and isotonic saline (placebo)infusion. The order of infusion is randomized. An interval of 30 minutes is planned between the two infusions.
  Interventions: Drug: remifentanil; Drug: placebo

INTERVENTIONS:
Drug: remifentanil — 0.05 mcg.kg-1.min-1 for 30 minutes by continuous endovenous infusion
Drug: placebo — NaCl 0.9 %

SUMMARY:
Sedation is widely used in mechanically ventilated patients. Propofol, benzodiazepines and opioids are the most used drugs. The study hypothesis is that sedation with remifentanil (an opioid drug) could improved respiratory pattern and effort in mechanically ventilated patients with rapid shallow breathing or high respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* pressure support ventilation or CPAP
* respiratory rate > 35.min-1
* respiratory rate/tidal volume > 105

Exclusion Criteria:

* vasoactive agents (dopamine lower than 5 mcg.kg-1.min-1 is not considered as vasoactive agent)
* body temperature > 38 °C
* Glasgow Coma Scale < 9
* FIO2 > 0.6
* PEEP > 10 cmH2O
* pH < 7.30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
respiratory rate/tidal volume | before and after remifentanil infusion; before and after placebo infusion.
pressure-time product | before and after remifentanil infusion; before and after placebo infusion.

SECONDARY OUTCOMES:
double product of respiratory system | before and after remifentanil infusion; before and after placebo infusion.
dynamic intrinsic PEEP | before and after remifentanil infusion; before and after placebo infusion.
adverse events | during all the study period
arterial pH | before and after remifentanil infusion; before and after placebo infusion.
level of sedation (RASS) | before and after remifentanil infusion; before and after placebo infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Natalini, MD, Principal Investigator — Fondazione Poliambulanza Istituto Ospedaliero
Locations (1):
- Intensive Care Unit, Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

REFERENCES:
- [Derived] Natalini G, Di Maio A, Rosano A, Ferretti P, Bertelli M, Bernardini A. Remifentanil improves breathing pattern and reduces inspiratory workload in tachypneic patients. Respir Care. 2011 Jun;56(6):827-33. doi: 10.4187/respcare.01014. Epub 2011 Feb 11. PMID 21333087